CLINICAL TRIAL: NCT03803111
Title: A Randomized Trial on Sequential Effects of Iron Therapy and Exercise Training in Patients With Heart Failure and Iron Deficiency
Brief Title: Effects of Iron Therapy and Exercise Training in Patients With Heart Failure and Iron Deficiency
Acronym: IronEx
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsoring and Screening of first patients was not sufficient
Sponsor: Herzzentrum Bremen (Other)
Responsible Party: Principal Investigator, Dr. Harm Wienbergen, Head of the Bremen Institute for Heart and Circulation Research (BIHKF), Herzzentrum Bremen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BIHKF-7162
Record Dates: First submitted 2019-01-08; First posted 2019-01-14 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Heart Failure With Reduced Ejection Fraction; Exercise Training; Ferric Carboxymaltose
Keywords: Heart Failure with Reduced Ejection Fraction; Exercise Training Program; Iron Deficiency
MeSH Terms: conditions — Iron Deficiencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Initial FCM (Experimental): Intravenous iron supplementation with FCM, subsequent (after 2 months) exercise training program
  Interventions: Drug: Initial FCM; Behavioral: Subsequent exercise training
- Initial exercise (Experimental): Exercise training program, subsequent (after 2 months) intravenous iron supplementation with FCM
  Interventions: Behavioral: Initial exercise training; Drug: Subsequent FCM

INTERVENTIONS:
Behavioral: Initial exercise training — Initial exercise training program
  Arms: Initial exercise
Drug: Initial FCM — Initial intravenous iron supplementation (FCM)
  Arms: Initial FCM
Drug: Subsequent FCM — Subsequent intravenous iron Supplementation (FCM) after 2 months
  Arms: Initial exercise
Behavioral: Subsequent exercise training — Subsequent exercise training program after 2 months
  Arms: Initial FCM

SUMMARY:
It is the aim of the study to prove, if intravenous supplementation with ferric carboxymaltose in iron-deficient patients with heart failure with reduced ejection fraction (HFrEF) leads to better exercise training effects compared to exercise training without previous iron supplementation.

DETAILED DESCRIPTION:
In patients with heart failure with reduced ejection fraction (HFrEF) exercise training (ET) is recommended. In iron-deficient HFrEF patients iron supplementation by ferric carboxymaltose (FCM) is recommended. Both treatment options (ET and iron supplementation) affect oxidative metabolism.

In this study iron-deficient HFrEF patients are included and randomly assigned to two study arms:

Study arm A: Intravenous iron supplementation with FCM, subsequent (after 2 months) ET program.

Study arm B: ET program, subsequent (after 2 months) intravenous iron supplementation with FCM.

Primary study endpoint is exercise capacity (Peak VO2). Secondary endpoints are 6-minute walking distance, NYHA class, echocardiographic parameters and the combined endpoint cardiovascular hospitalizations and death.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure with reduced ejection fraction ≤ 40%
* New York Heart Failure Asssociation class II-III
* Iron deficiency (ferritin < 100 ng/ml or 100-299 ng/ml, if transferrin saturation < 20%)

Exclusion Criteria:

* Planned cardiovascular interventions (such as bypass surgery or valve interventions)
* Acute coronary Syndrome
* Malignant rhythm disturbances
* Acute or chronic infection
* Reduced prognosis or exercise capacity by non-cardiac comorbidities
* Missing informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Exercise capacity (Peak VO2) | Change from baseline to 4 months
  Peak VO2 is measured by spiroergometry

SECONDARY OUTCOMES:
6 Minute walking distance | Change from baseline to 4 months
  To further assess exercise capacity
New York Heart Association class (class I, II, III, IV with class I = best status, and class IV = worst status) | Improvement or deterioration of NYHA class from baseline to 4 months
  To assess symptoms
Echocardiographic ejection fraction of left ventricular function (measured in %, the lower the worse) | Improvement or deterioration of ejection fraction from baseline to 4 months
  Systolic and diastolic function, chamber diameters, strain analyses
Combined endpoint cardiovascular hospitalizations and death | After 2 and 4 months
  To assess major events

CONTACTS AND LOCATIONS:
Locations (1):
- Bremer Institut für Herz- und Kreislaufforschung, Bremen, Germany